CLINICAL TRIAL: NCT07296601
Title: Expert Consensus on the Clinical Use of Skin Boosters: A Delphi-Based Recommendation Framework
Status: Enrolling by invitation | Type: Observational
Sponsor: Venus Research Center (Other)
Responsible Party: Sponsor
Other Study IDs: Skin Booster-VenusRC
Record Dates: First submitted 2025-12-08; First posted 2025-12-22 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Aesthetic Procedures; Cosmetic Techniques; Skin Ageing
Keywords: Skin booster; rejuvenation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Expert Panel: A cohort of dermatology and aesthetic medicine experts participating in a Modified Delphi process to develop consensus recommendations on skin booster use.

SUMMARY:
This consensus research project aims to develop standardized, evidence-based recommendations for the clinical use of skin boosters in aesthetic dermatology. Despite their widespread adoption for improving skin hydration, texture, and dermal quality, current practice patterns vary significantly across clinicians and regions, with limited unified guidelines. Using a structured Delphi methodology, the study will gather expert opinions from dermatologists and aesthetic medicine specialists to achieve agreement on key aspects of skin booster therapy, including indications, patient selection, injection techniques, dosing protocols, product selection, treatment intervals, expected outcomes, and safety considerations.

The project seeks to establish practical, consensus-driven guidelines that can harmonize clinical practice, enhance treatment outcomes, and ensure patient safety. The final recommendations will serve as a reference framework for practitioners and contribute to the standardization of skin quality enhancement treatments.

DETAILED DESCRIPTION:
Skin boosters have become an increasingly popular modality in aesthetic dermatology due to their ability to enhance skin hydration, elasticity, texture, and overall dermal quality through minimally invasive intradermal injections. Despite their rapid integration into clinical practice, current approaches to skin booster therapy remain highly variable. Differences exist in product selection, injection depth, dosing regimens, treatment intervals, technique, indications, and safety monitoring. Moreover, the evidence base is still evolving, and most available data come from fragmented clinical studies or manufacturer-driven guidelines. As a result, there is a significant need for unified, expert-driven recommendations that can standardize practice, optimize patient outcomes, and minimize complications.

This research project aims to develop comprehensive, evidence-informed consensus guidelines for the use of skin boosters in aesthetic practice. The study will use a structured Delphi methodology to gather and synthesize the perspectives of leading dermatologists and aesthetic medicine specialists. Through multiple iterative rounds, experts will evaluate and rate a series of statements addressing key clinical domains including: appropriate indications; patient selection criteria; anatomical considerations; recommended injection depths and techniques; dosing strategies; frequency and number of treatment sessions; choice of products (e.g., HA-based, polynucleotides, bio-remodeling agents); combination therapies; expected outcomes; management of adverse events; and contraindications.

The consensus-building process ensures anonymity, reduces bias, and encourages equal participation among experts. Quantitative analyses (e.g., percentage agreement thresholds, median and interquartile range scoring) will be used to determine which statements achieve consensus. Statements not reaching agreement will be revised and re-evaluated in subsequent rounds until final consensus is achieved.

By the end of the project, the expert panel will produce clear, standardized, and clinically actionable recommendations that can be used globally or regionally to harmonize the use of skin boosters. These guidelines will support clinicians by improving the consistency and quality of care, informing training programs, guiding patient counseling, and reducing complication rates. Ultimately, the project aims to fill a critical gap in aesthetic dermatology literature by establishing a scientifically grounded, consensus-driven framework for safe and effective skin booster therapy

ELIGIBILITY:
Inclusion Criteria:

* Inclusion Criteria

Experts will be eligible to participate if they meet all of the following:

Board-certified dermatologist or aesthetic physician

With recognized qualification in dermatology, aesthetic medicine, plastic surgery, or related fields.

Minimum clinical experience

At least 5 years of experience performing aesthetic injectable procedures.

OR at least 3 years of consistent use of skin boosters in clinical practice.

Demonstrated expertise in skin booster therapy

Must have performed ≥100 skin booster procedures overall,

OR ≥20 sessions per year over the past 2 years.

Active clinical practice

Currently practicing in an aesthetic or dermatology clinic, medical center, or hospital.

Authorship or contribution to aesthetic/dermatology education (desirable but not mandatory)

Publications, lectures, workshop instruction, or conference involvement in aesthetics.

Ability to participate in Delphi rounds

Must agree to complete all survey rounds within the specified timeframe.

Must be fluent in the language used for the study (e.g., English or Arabic).

Willingness to provide informed consent

Voluntary participation with confidentiality maintained.

Exclusion Criteria:

* Less than the required experience

<5 years of aesthetic practice

OR insufficient hands-on experience with skin booster injections.

Limited familiarity with skin booster products or techniques

No regular use in the last 2 years.

Has not performed the minimum number of required procedures.

Industry conflict of interest

Direct employment by a company manufacturing skin booster products.

Significant financial relationship with a single product manufacturer that may bias responses.

Inability to commit to multiple Delphi rounds

Anticipated non-compliance or non-response in iterative rounds.

Non-clinical or administrative professionals

Those not actively practicing (e.g., retired, research-only positions, students, trainees).

Participation in a competing guideline project

Experts currently serving on another skin booster consensus panel to avoid duplication or bias.

Failure to provide informed consent

Declines participation or withdraws consent at any time.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population will consist of a purposively selected panel of experts in aesthetic dermatology and skin booster therapy. Participants will include board-certified dermatologists, aesthetic physicians, and plastic surgeons with substantial clinical experience in administering injectable skin quality treatments. The expert panel will represent a diverse range of clinical backgrounds, geographical regions, and practice settings to ensure comprehensive and balanced perspectives.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2025-12-25 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Degree of Consensus on Clinical Recommendations | 6-12 weeks
  1. Degree of Consensus on Clinical Recommendations
     Definition: The level of expert agreement on each statement related to skin booster therapy.
     Measurement Method:
     Likert scale ratings (e.g., 1-9).
     Consensus threshold often defined as:
     ≥75% agreement within the 7-9 range (agreement)
     ≤15% ratings in the 1-3 range (disagreement)
     Outcome: Identification of statements that meet consensus criteria for inclusion in the final guideline.
  2. Development of Final Consensus Guidelines
  Definition: The creation of a unified, evidence-informed set of recommendations on skin booster use.
  Measurement Method:
  Number of statements that reach consensus across all Delphi rounds.
  Completeness of guideline domains (indications, technique, dosing, safety, etc.).
  Outcome: A finalized recommendations document for clinicians.

SECONDARY OUTCOMES:
Implementation Readiness of Final Recommendations | 6-12 weeks
  Definition: Practicality and ease of applying the guidelines in real-world clinical settings.
  Measurement Method:
  Expert evaluation of feasibility (Likert scale).
  Assessment of clarity and actionability of statements.
  Outcome: Determines how applicable the recommendations are in routine practice.

CONTACTS AND LOCATIONS:
Locations (1):
- Venus Research Center, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No
Delphi studies do not collect patient data, medical records, biological samples, or identifiable clinical information. Experts only give opinions, not "IPD." Their responses are anonymized, and sharing identifiable expert-level responses is not required and often discouraged